CLINICAL TRIAL: NCT01019148
Title: Characteristics of Patients With Recessive Dystrophic Epidermolysis Bullosa
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jean Yuh Tang, Professor, Stanford University
Other Study IDs: SU-11182009-4402
Record Dates: First submitted 2009-11-20; First posted 2009-11-25 (Estimated); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Epidermolysis Bullosa Dystrophica
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsies, serum

SUMMARY:
Recessive dystrophic epidermolysis bullosa (RDEB) is a disease caused by genetic mutations in the gene for type VII collagen. Patients with RDEB develop large, severely painful blisters and open wounds from minor trauma to their skin. We are screening subjects with RDEB to evaluate characteristics of the subjects and their cells in order to develop new strategies of therapy and determine whether subjects could be candidates for treatment studies.

DETAILED DESCRIPTION:
We will obtain a detailed medical history and will perform a skin examination and brief physical exam. Photographs may be taken. We will ask questions about the size and duration wounds.

LAB TESTS We will draw blood to determine overall health status to include Hepatitis B, Hepatitis C, and Human Immunodeficiency Virus (HIV) testing. Genetic testing may also be performed.

BIOPSIES Biopsies may be collected to check for Collagen 7 and for antibodies to Collagen 7.

Based on the results obtained, it may be possible to identify patients who would qualify to participate in current or future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of RDEB by local dermatologist
* 7 years of age or older

Exclusion Criteria:

-Medical instability limiting ability to travel to Stanford University Medical Center

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with RDEB by a local dermatologist who are medically stable enough to travel to Stanford University Medical Center. Patients should also be at least 7 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2009-11-10 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of subjects with Recessive Dystrophic Epidermolysis Bullosa | 10 years
  Identification of subjects with Recessive Dystrophic Epidermolysis Bullosa for future studies

CONTACTS AND LOCATIONS:
Overall Officials: Jean Tang, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States